CLINICAL TRIAL: NCT04072289
Title: SMILE (Small Incision Lenticule Extraction) in the DoD (Department of Defense)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Principal Investigator, John Cason, Principle Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD-2016.0055
Record Dates: First submitted 2019-03-11; First posted 2019-08-28 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Myopia; Astigmatism
Keywords: refractive surgery; small incision lenticule extraction; femtosecond laser; myopia; astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: comparative cohort trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Low cylinder (treatment) (Experimental): 0.25D and 0.50D cylinder treatments will be measured and treated by the laser.
  Interventions: Device: Visumax spherocylindrical treatment
- Low cylinder (no treatment) (No Intervention): 0.25D and 0.50D cylinder treatments will be measured but not treated by the laser. No spherical equivalent will be used.

INTERVENTIONS:
Device: Visumax spherocylindrical treatment — treatment of low cylinder (<0.75D)
  Arms: Low cylinder (treatment)

SUMMARY:
The Use of the VisuMaxTM Femtosecond Laser Small-Incision Lenticule Extraction (SMILE) Procedure for the Correction of Myopia with or without Astigmatism study is a prospective, non-randomized, multicenter clinical study that will be conducted by the Navy Refractive Surgery Center, Naval Medical Center San Diego, CA in collaboration with the U.S. Air Force 59th Medical Wing, Wilford Hall Eye Center, TX, and the U.S. Army Warfighter Refractive Eye Surgery Program and Research Center, Fort Belvoir Community Hospital, VA.

DETAILED DESCRIPTION:
Prospective, multicenter, open-label, non-randomized clinical trial with bilateral commercial treatment for FDA approved indications and unilateral treatments for investigational refractive errors. Data from each treated eye of subjects will be treated independently. Monovision treatments and retreatments of the study eye will not be allowed during the course of the study. Successful bilateral treatment is required for performance based testing and patient reported outcome testing. Subjects will be randomized into the 0.25 and 0.50 sphere only and spherical cylinder bins using a sequential alternating randomization with an equal number assigned to both bins. Other subjects will be assigned to the bins they qualify for as they are enrolled into the study. Appointments are given to patients requesting refractive surgery randomly.

Three military sites in the U.S.A.: Navy Refractive Surgery Center, Naval Medical Center San Diego, CA in collaboration with the U.S. Air Force 59th Medical Wing, Wilford Hall Eye Center, TX, and the U.S. Army Warfighter Refractive Eye Surgery Program and Research Center, Fort Belvoir Community Hospital, VA.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 22 years of age and older either active duty or dependents who are eligible for care;
2. Myopia from ≥ 0 D to ≤ -10.00 D with ≤ -3.00 D cylinder and MRSE ≥ -1.00 D to

   ≤ -11.50 D in the eye(s) to be treated;
3. A stable refraction for the past year, as demonstrated by a change in MRSE of ≤ 0.50 D in the eyes to be treated;
4. A difference between cycloplegic and manifest refractions of

   ≤ 0.75 D spherical equivalent in both eye(s);
5. UCVA 2 lines worse than BCVA in the treated eye(s);
6. BSCVA at least 20/20 in the treated eye(s);
7. Discontinue use of contact lenses for at least 4 weeks (for hard lenses) or 2 weeks (for soft lenses) prior to the preoperative examination, and through entire study. The subject shall not be considered a contact lens wearer if they are not wearing hard contact lenses for 4 weeks or soft contact lenses for 2 weeks.
8. All contact lens wearers must demonstrate a stable refraction (within ±0.5 D), as determined by MRSE, on two consecutive examinations at least 7 days apart, in the eye(s) to be treated;
9. Central corneal thickness of at least 500 microns in the both eye(s);
10. Willing and able to return for scheduled follow-up examinations;
11. Able to provide written informed consent and follow study instructions in English.
12. Permission of the Commanding Officer for active duty subjects to receive refractive surgery and participate in the study.

Exclusion Criteria:

1. Manifest cylinder of more than -3.00 D;
2. Estimated treatment depth is less than 250 microns from the corneal endothelium;
3. Eye to be treated is targeted for monovision;
4. Keratometry readings via Sim-K values less than 40.00 D;
5. Abnormal corneal topographic findings, e.g. keratoconus, pellucid marginal degeneration in either eye;
6. History of or current anterior segment pathology, including cataracts in the eye to be treated;
7. Clinically significant dry eye syndrome unresolved by treatment in either eye;
8. Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease in the either eye;
9. Ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect) in either eye;
10. Irregular or unstable (distorted/not clear) corneal mires on central keratometry images in either eye;
11. History of ocular herpes zoster or herpes simplex keratitis;
12. Deep orbits, strong blink, anxiety, pterygium, or any other finding suggesting difficulty in achieving or maintaining suction;
13. Difficulty following directions or unable to fixate;
14. Previous intraocular or corneal surgery of any kind in the eye to be treated, including any type of surgery for either refractive or therapeutic purposes;
15. History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP > 21 mmHg in either eye;
16. History of diabetes, diagnosed autoimmune disease, connective tissue disease or clinically significant atopic syndrome;
17. Immunocompromised or requires chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing;
18. History of known sensitivity to planned study medications;
19. Participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation;
20. Pregnant or lactating;
21. Anyone who has the potential to deploy or relocate during the follow-up period.
22. Systemic Medications that may confound the outcome of the study or increase risk to the subject, including but not limited to steroids, antimetabolites, etc.
23. Evidence of retinal vascular disease.
24. Glaucoma suspects by exam findings or family history.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Measured postoperative refractive sphere and cylinder | 12 months
  manifest refraction spherical equivalent and manifest refractive cylinder refraction
Measured distance visual acuity | 12 months
  uncorrected visual acuity of 20/40 or better

SECONDARY OUTCOMES:
Measured difference in manifest refraction between 2 postoperative visits | latter of 2 postoperative refractions performed at least 3 months apart or at 3 months after surgery when compared with the 1 month interval
  95% of eyes <1.00D of MRSE change at latter of 2 postop refractions
Calculated rate of change in manifest refraction | latter of 2 postoperative refractions performed at least 3 months apart or at 3 months after surgery when compared with the 1 month interval
  mean rate of change of MRSE <0.5D/year (0.04D/mo)
Calculated decreased rate of change in manifest refraction | latter of 2 postoperative refractions performed at least 3 months apart or at 3 months after surgery when compared with the 1 month interval
  mean rate of change of MRSE decreases monotonically over time
Calculated stable rate of change in manifest refraction | latter of 2 postoperative refractions performed at least 3 months apart or at 3 months after surgery when compared with the 1 month interval
  95% CI for the mean rate of change includes zero
Measured best corrected visual acuity (method 1) | 12 months
  incidence of best spectacled correction worse than 20/40
Measured best corrected visual acuity (method 2) | 12 months
  incidence of loss of >2 lines of best spectacled corrected visual acuity
Measured refractive cylinder | 12 months
  incidence of induced cylinder >2D
Incidence of adverse events | 12 months
  incidence of adverse events
Incidence of patient reported visual phenomena | 12 months
  incidence of patient subjective symptoms
Measured contrast sensitivity | 12 months
  change in contrast sensitivity from preop to postop

CONTACTS AND LOCATIONS:
Overall Officials: John B. Cason, M.D., Principal Investigator — United States Naval Medical Center, San Diego; Matthew C. Caldwell, M.D., Principal Investigator — Wilford Hall Air Force Hospital; Bruce A Rivers, M.D., Principal Investigator — Ft. Belvoir Army Hospital
Locations (1):
- Navy Warfighter Refractive Surgery Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with Zeiss Meditech by Data Sharing Agreement and with the FDA